CLINICAL TRIAL: NCT06766773
Title: Warming with a Composite Warming Strategy Reduces Intraoperative Hypothermia in Patients Undergoing Open Hepatectomy for Liver Cancer: a Randomized Controlled Study
Brief Title: Composite Warming Strategy Reduces Intraoperative Hypothermia in Open Hepatectomy for Liver Cancer
Acronym: CWSRIH-HCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Neijiang (Other)
Responsible Party: Principal Investigator, Ou Jiang, Director of Cancer Center, The First People's Hospital of Neijiang
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-lunshenpi-32
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HCC
Keywords: Intraoperative hypothermia; Open hepatectomy for liver cancer; Composite warming strategy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: perioperative mandatory warming measures (Placebo Comparator)
  Interventions: Procedure: perioperative mandatory warming measures
- Compound heating strategy (Experimental)
  Interventions: Procedure: Compound heating strategy

INTERVENTIONS:
Procedure: Compound heating strategy — After the surgery begins, a temperature monitoring device (disposable medical temperature sensor provided by the limited company) is inserted into the patient's nasopharynx to record the core temperature, while activating the water blanket and forced air heating system.
  Arms: Compound heating strategy
Procedure: perioperative mandatory warming measures — perioperative mandatory warming measures
  Arms: Control group: perioperative mandatory warming measures

SUMMARY:
The composite warming strategy has a certain effect on preventing hypothermia during cancer liver resection surgery. This study aims to explore the application of compound warming strategy in perioperative nursing of cancer liver resection.

This study will compare two groups: the control group using perioperative forced warming measures, and the experimental group using a composite warming strategy.

Main objective: Intraoperative temperature changes Secondary objective: incidence of complications The investigators' investigated the practicality and effectiveness of a combined warming strategy in open liver resection surgery. In addition, the investigators also conducted a quantitative correlation study on the incidence of hypothermia during the surgical process. This provides evidence-based guidance for the prevention of hypothermia during surgery.

DETAILED DESCRIPTION:
Research Title: Warming with a Composite Warming Strategy Reduces Intraoperative Hypothermia in Patients Undergoing Open Hepatectomy for Liver Cancer: A Randomized Controlled Study Background: Perioperative hypothermia is a clinical condition characterized by a core body temperature dropping below 36 ° C during the perioperative period, which is a common complication in anesthesia and open abdominal surgery. This state can lead to various perioperative complications, including but not limited to surgical site infections, arrhythmia, and cardiac obstruction.

Main objective: Intraoperative temperature changes Secondary objective: incidence of complications Meaning:The investigators' investigated the practicality and effectiveness of a combined warming strategy in open liver resection surgery. In addition, the investigators also conducted a quantitative correlation study on the incidence of hypothermia during the surgical process. This provides evidence-based guidance for the prevention of hypothermia during surgery. In addition, the investigators also conducted a quantitative correlation study on the incidence of hypothermia during the surgical process.

Innovation: The innovation of this article lies in the first verification of the practicality and effectiveness of the composite warming strategy in open liver resection surgery.

Expected outcome: The practical and effective use of a combined warming strategy in open liver resection surgery. In terms of anesthesia duration, blood loss, fluid replacement, and PACU observation duration, the composite warming strategy may have better results than the forced air warming system.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years.
* Scheduled for elective open hepatectomy to treat hepatocellular carcinoma, confirmed by preoperative biopsy or imaging.
* Adequate liver function (Child-Pugh score A or B).
* American Society of Anesthesiologists (ASA) physical status classification of I, II, or well-controlled III.
* Informed consent provided for participation.

Exclusion Criteria:

* Aged under 18 or over 75 years.
* Metastatic liver disease or emergency liver surgery required.
* Chronic analgesic use that could interfere with pain assessment.
* Participation in another clinical trial within the past 30 days.
* Contraindications to warming devices (e.g., certain skin conditions or advanced peripheral vascular disease).
* Pregnant or lactating.
* Presence of an implantable device (e.g., pacemakers or defibrillators) that could be affected by warming strategies.
* Cognitive impairment or psychiatric disorders affecting study understanding or informed consent.
* Use of medications/substances impacting thermoregulation (e.g., illicit drugs, alcohol abuse, antipyretics).
* History of malignancies other than liver cancer affecting survival or perioperative risk.
* Recent history (within six months) of myocardial infarction or cerebrovascular accident.
* Uncontrolled diabetes mellitus or other significant endocrine disorders.
* Severe anemia (hemoglobin below a predetermined threshold).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative temperature changes | At the beginning of the surgery; every 5 minutes during surgery; after the surgery is completed.
  Intraoperative temperature changes: After the surgery begins, a temperature monitoring device (disposable medical temperature sensor provided by the limited company) is inserted into the patient's nasopharynx to record the core temperature, while activating the water blanket and forced air.

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Neijiang, Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] John M, Ford J, Harper M. Peri-operative warming devices: performance and clinical application. Anaesthesia. 2014 Jun;69(6):623-38. doi: 10.1111/anae.12626. Epub 2014 Apr 10. PMID 24720346
- [Background] Andrzejowski J, Hoyle J, Eapen G, Turnbull D. Effect of prewarming on post-induction core temperature and the incidence of inadvertent perioperative hypothermia in patients undergoing general anaesthesia. Br J Anaesth. 2008 Nov;101(5):627-31. doi: 10.1093/bja/aen272. Epub 2008 Sep 26. PMID 18820248
- [Background] Kvolik S, Jukic M, Matijevic M, Marjanovic K, Glavas-Obrovac L. An overview of coagulation disorders in cancer patients. Surg Oncol. 2010 Mar;19(1):e33-46. doi: 10.1016/j.suronc.2009.03.008. Epub 2009 Apr 25. PMID 19394816
- [Background] Kanikarla Marie P, Fowlkes NW, Afshar-Kharghan V, Martch SL, Sorokin A, Shen JP, Morris VK, Dasari A, You N, Sood AK, Overman MJ, Kopetz S, Menter DG. The Provocative Roles of Platelets in Liver Disease and Cancer. Front Oncol. 2021 Jul 21;11:643815. doi: 10.3389/fonc.2021.643815. eCollection 2021. PMID 34367949
- [Background] Staikou C, Paraskeva A, Drakos E, Anastassopoulou I, Papaioannou E, Donta I, Kontos M. Impact of graded hypothermia on coagulation and fibrinolysis. J Surg Res. 2011 May 1;167(1):125-30. doi: 10.1016/j.jss.2009.07.037. Epub 2009 Aug 26. PMID 19932906
- [Background] Birgin E, Kaslow SR, Hetjens S, Correa-Gallego C, Rahbari NN. Minimally Invasive versus Open Liver Resection for Stage I/II Hepatocellular Carcinoma. Cancers (Basel). 2021 Sep 25;13(19):4800. doi: 10.3390/cancers13194800. PMID 34638285
- [Background] Xu H, Xu G, Ren C, Liu L, Wei L. Effect of forced-air warming system in prevention of postoperative hypothermia in elderly patients: A Prospective controlled trial. Medicine (Baltimore). 2019 May;98(22):e15895. doi: 10.1097/MD.0000000000015895. PMID 31145350
- [Background] Simegn GD, Bayable SD, Fetene MB. Prevention and management of perioperative hypothermia in adult elective surgical patients: A systematic review. Ann Med Surg (Lond). 2021 Nov 14;72:103059. doi: 10.1016/j.amsu.2021.103059. eCollection 2021 Dec. PMID 34840773
- [Background] Diaz M, Becker DE. Thermoregulation: physiological and clinical considerations during sedation and general anesthesia. Anesth Prog. 2010 Spring;57(1):25-32; quiz 33-4. doi: 10.2344/0003-3006-57.1.25. PMID 20331336
- [Background] Balki I, Khan JS, Staibano P, Duceppe E, Bessissow A, Sloan EN, Morley EE, Thompson AN, Devereaux B, Rojas C, Rojas C, Siddiqui N, Sessler DI, Devereaux PJ. Effect of Perioperative Active Body Surface Warming Systems on Analgesic and Clinical Outcomes: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2020 Nov;131(5):1430-1443. doi: 10.1213/ANE.0000000000005145. PMID 33079867
- [Derived] Yi N, Wang Z, Cui R. Warming with a composite warming strategy reduces intraoperative hypothermia in patients undergoing open hepatectomy for liver cancer: A randomized controlled study. Medicine (Baltimore). 2025 Feb 21;104(8):e41616. doi: 10.1097/MD.0000000000041616. PMID 39993117